CLINICAL TRIAL: NCT02408666
Title: EEG@HOME (Phase 1 of the Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Pilipili NV (Industry); Imec (Industry)
Responsible Party: Principal Investigator, Neurologie, Prof. dr. Kristl Vonck, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2014/0319
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interview (Other): Interview of epilepsy patients and their family about their experience with epilepsy, EEG registrations and daily life.
  Interview of EEG-technologists and neurologists about their experience with EEG registrations and expections when thinking of a ideal EEG-cap.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview

SUMMARY:
The goal of this project is the development of an EEG-cap (min. 21 electrodes) with user-friendly active dry electrodes that meets the expectations of the users regarding comfort and esthetics, without losing sight of the functional and technical demands for recording high quality EEG signals. The purpose is to use the EEG-cap to investigate clinical neurological disorders (e.g. epilepsy). The EEG-cap could also be used at home so that hospital admission in the EMU can be avoided for some patients and an increasing number of patients can be examined.

In Phase 1 of the project epilepsy patients and their family will be interviewed about their personal experiences with the condition, EEG registrations, daily life, ... . In addition EEG-technologists and neurologists will be interviewed about their experience with EEG registrations and what features their dream EEG-cap would have. The purpose is to gain insight in the wishes and expectations of the end users so we can take this into account when designing of the EEG-cap. This interview is anticipated to take approximately 1 hour.

Minimum 5 - maximum 50 patients and their family will be interviewed. Minimum 5 - maximum 50 EEG-technologists or neurologists will be interviewed.

The results of the interviews will be analysed by the design company pilipili nv.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy patient or EEG-technologist or neurologist

Exclusion Criteria:

* No experience with EEG

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
User wishes and expectations (questionnaire) | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium